CLINICAL TRIAL: NCT00152243
Title: A Randomized Controlled Study of Postoperative Adjuvant Chemotherapy of UFT Compared With Surgery Alone for Serosa-negative Advanced Gastric Cancer (NSAS-GC)
Brief Title: A Randomized Controlled Study of Postoperative Adjuvant Chemotherapy of Uracil- Tegafur (UFT) Compared With Surgery Alone (NSAS-GC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taiho Pharmaceutical Co., Ltd., Taiho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01023003
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Gastric Cancer
Keywords: Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Tegafur; Uracil; Surgical Procedures, Operative

ARMS (2):
- 1 (Experimental): UFT (uracil, tegafur)
  Interventions: Drug: UFT (uracil, tegafur)
- 2 (Other): Surgery alone
  Interventions: Procedure: Surgery alone

INTERVENTIONS:
Drug: UFT (uracil, tegafur) — uracil-tegafur 360 mg per square meter per day orally 16 months
  Arms: 1
Procedure: Surgery alone — Gastrectomy of tumour node metastasis(TNM) stage T2N1-2 gastric cancer.
  Arms: 2

SUMMARY:
This is a controlled study designed to evaluate the efficacy of UFT on survival compared with surgery alone. Patients will be randomly assigned to receive either surgery alone or surgery followed by UFT within 6 weeks after curative resection. To assess treatment response, data on recurrence and survival will be collected for 5 years after enrollment of the last patient. To evaluate safety, data on adverse events will be collected for 16 months after the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 75
* Performance status 0 , 1, or 2 (ECOG)
* Hematopoietic WBC ≥ 4,000/mm^3 Platelet ≥ 100,000/mm^3
* Hepatic AST and ALT ≤ 2 times upper limit of normal(ULN) Total bilirubin ≤ 1.5 times ULN
* Renal BUN ≤1.5 times ULN Creatinine ≤ 1.5 times ULN

Exclusion Criteria:

* Prior anticancer treatment

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 1997-06; Primary Completion 2006-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Overall survival and relapse-free survival | every course for first three courses, then every other course

SECONDARY OUTCOMES:
Adverse events | any time

CONTACTS AND LOCATIONS:
Overall Officials: Toshifusa Nakajima, MD, Principal Investigator — Cancer Institute Hospital
Locations (1):
- Cancer Institute Hospital, Japanese Foundation for Cancer Research, 3-10-6, Ariake, Koto-ku, Tokyo, Japan

REFERENCES:
- [Result] Nakajima T, Kinoshita T, Nashimoto A, Sairenji M, Yamaguchi T, Sakamoto J, Fujiya T, Inada T, Sasako M, Ohashi Y; National Surgical Adjuvant Study of Gastric Cancer Group. Randomized controlled trial of adjuvant uracil-tegafur versus surgery alone for serosa-negative, locally advanced gastric cancer. Br J Surg. 2007 Dec;94(12):1468-76. doi: 10.1002/bjs.5996. PMID 17948223